CLINICAL TRIAL: NCT04894591
Title: Jazz Emerge 402: Phase IV Observational Study to Collect Safety and Outcome Data in Real-World Setting in Adult Patients With Extensive Stage Small Cell Lung Cancer (SCLC) Receiving Zepzelca
Brief Title: To Assess the Effectiveness and Safety of Zepzelca in Adult Patients With Extensive Stage Small Cell Lung Cancer (SCLC)
Acronym: SCLC
Status: Completed | Type: Observational
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: JZP712-402
Record Dates: First submitted 2021-04-30; First posted 2021-05-20 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Extensive-stage Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — PM 01183

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Zepzelca — Zepzelca is administered by intravenous infusion over 60 minutes every 21 days. Date, dose prescribed and received will be collected at each Zepzelca infusion.
  Other Names: lurbinectedin

SUMMARY:
To assess the effectiveness and safety of Zepzelca in adult participants with extensive stage small cell lung cancer (SCLC) in real-world clinical practice.

DETAILED DESCRIPTION:
A phase IV, prospective, single arm, multi-center, observational study to collect safety and outcome data of Zepzelca in adult participants with extensive stage SCLC previously exposed to at least one line of treatment with platinum-based chemotherapy. Patients enrolled in the study will be encouraged to complete patient reported outcome (PRO) questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has initiated or will be receiving Zepzelca treatment in line with the local Zepzelca prescribing information.
2. Decision to initiate treatment with Zepzelca was made as per investigator's routine treatment practice prior to enrollment in the study.
3. Patient, or a legally acceptable representative, signed the informed consent before any study-related activities are undertaken.
4. Patients initiating Zepzelca treatment in second-line.
5. Patients who are sensitive to platinum-based chemotherapy with CTFI≥180 days. The CTFI is defined as the length of time from last platinum dose to time of relapse or disease progression.
6. Eastern Cooperative Oncology Group performance status (ECOG) ≤1

Exclusion Criteria:

1. Patients who discontinued a prior Zepzelca treatment due to adverse events.
2. Patient who received more than 2 cycles of Zepzelca treatment in their current treatment schedule.
3. Patient received treatment with any investigational agent within 30 days prior to first Zepzelca infusion or plans to use another investigational agent while receiving Zepzelca.
4. Known CNS involvement prior to Zepzelca treatment.
5. Patients who were treated with Zepzelca in later lines rather than in second-line treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with extensive SCLC treated with Zepzelca.
Sampling Method: Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | up to 6 months after first infusion

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 6 months after first infusion
Progression-Free Survival (PFS) | up to 6 months after first infusion
Duration of Response (DoR) | up to 6 months after first infusion
Disease Control Rate (DCR) | up to 6 months after first infusion
Distribution of Treatment Patterns in Participants Measured by Number of Days in a Cycle, Dose Intensity, Number of Dose Reductions and Dose Delays, Number of Cycles Summarized by Number of Previous Lines of Therapy | up to 6 months after first infusion
Assessing Safety and Tolerability of Zepzelca by Assessing the Number of Participants with Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESI) | up to 6 months after first infusion
Time to Response to Zepzelca | up to 6 months after first infusion
Participants Health-related Quality of Life (HRQOL) using Patient Reported Outcome (PRO) Questionnaires | up to 6 months after first infusion
Overall Survival (OS) in Other Subgroups of Interest | up to 6 months after first infusion
Progression-Free Survival (PFS) in Other Subgroups of Interest | up to 6 months after first infusion
Duration of Response (DoR) in Other Subgroups of Interest | up to 6 months after first infusion
Disease Control Rate (DCR) in Other Subgroups of Interest | up to 6 months after first infusion
Assessing Safety and Tolerability of Zepzelca by Assessing the Number of Participants with SAEs and AESI in Subgroups of Interest | up to 6 months after first infusion

CONTACTS AND LOCATIONS:
Locations (41):
- United States (32):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Eastern Connecticut Hematology and Oncology, Norwich, Connecticut
  - ASCLEPES Research Centers, Brooksville, Florida
  - Woodlands Medical Specialists - Woodlands Center For Specialized Medicine, Pensacola, Florida
  - Mid-Illinois Hematology & Oncology Associates, Normal, Illinois
  - Goshen Health Center for Cancer Care, Goshen, Indiana
  - Siouxland Regional Cancer Center dba June E. Nylen Cancer Center, Sioux City, Iowa
  - Stormont-Vail Cancer Center-Stormont-Vail Healthcare - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Pikeville Medical Center - Leonard Lawson Cancer Center, Pikeville, Kentucky
  - West Jefferson Cancer Center, Marrero, Louisiana
  - MMCORC - HealthPartners Institute, Saint Louis Park, Minnesota
  - Singing River Health System, Pascagoula, Mississippi
  - Central Care Cancer Center, Bolivar, Missouri
  - Benefis Medical Group, Great Falls, Montana
  - Regional Cancer Care Associates LLC (RCCA), Hackensack, New Jersey
  - Center for Clinical Research-Rochester General Hospital, Rochester, New York
  - Montefiore Medical Center (MMC) - Montefiore Medical Park (MMP), The Bronx, New York
  - University of North Carolina NASH Cancer Center, Rocky Mount, North Carolina
  - Trinity Cancercare Center, Minot, North Dakota
  - Gabrail Cancer Center Research, Canton, Ohio
  - Tri-County Hematology & Oncology Associates, Inc, Massillon, Ohio
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - Charleston Hematology Oncology Associates, PA, Charleston, South Carolina
  - Carolina Blood & Cancer Care Associates, Rock Hill, South Carolina
  - Lexington Oncology Associates, West Columbia, South Carolina
  - Monument Health Cancer Care Institute, Rapid City, South Dakota
  - Baptist Cancer Center, Memphis, Tennessee
  - Baylor Scott & White Medical Center - Temple, Temple, Texas
  - Tranquil Clinical Research, Webster, Texas
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
- Canada (9):
  - Cape Breton Cancer Centre, Sydney, Nova Scotia
  - Southlake Regional Health Centre (York County Hospital), Newmarket, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Integre Universitaire de Sante et de Services Sociaux du Saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - Centre integre de sante et de services sociaux de Chaudiere-Appalaches, Lévis, Quebec
  - Centre integre de Sante Et De Services Sociaux du Bas-Saint-Laurent Hopital regional de Rimousk, Rimouski, Quebec
  - Universite Laval - Institut Universitaire de Cardiologie et de Pneumologie de Quebec (IUCPQ) (Hopital Laval), Sainte-Foy, Quebec
  - CIUSSS de L'Estrie - CHUS - Hopital Fleurimont, Sherbrooke, Quebec